CLINICAL TRIAL: NCT04240249
Title: Constructive Self Assertiveness Via the Internet
Acronym: R2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Responsible Party: Principal Investigator, Per Carlbring, Professor, Stockholm University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Respect
Record Dates: First submitted 2020-01-15; First posted 2020-01-27 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Problems With Self-assertiveness

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with three groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Constructive self-assertiveness with guidance (Experimental): 10 weeks of internet-based treatment with weekly assignments. The homework is commented on by the guide using electronic communication.
  Interventions: Behavioral: Constructive self-assertiveness program via the internet
- Constructive self-assertiveness without guidance (Experimental): 10 weeks of internet-based treatment with weekly assignments. The homework is NOT commented on by any guide. Hence, same treatment as group 1 but without guidance.
  Interventions: Behavioral: Constructive self-assertiveness program via the internet
- Waitlist control (No Intervention): No treatment, no guidance, just waiting for 10 weeks. After the ten weeks the participants will receive the treatment.

INTERVENTIONS:
Behavioral: Constructive self-assertiveness program via the internet — Participants will get one "chapter" a week to work with. All chapters are presented on web pages and include information and exercises and end with homework assignments.
  Arms: Constructive self-assertiveness with guidance; Constructive self-assertiveness without guidance

SUMMARY:
Some people have problems with self-assertiveness. That can have negative impact on their lives. This study will test a constructive self-assertiveness intervention program delivered online. In addition, the relative effect of guidance during the intervention will be investigated.

In a randomized controlled trial three groups will be compared:

1. constructive self-assertiveness with guidance
2. constructive self-assertiveness without guidance
3. Waitlist control

DETAILED DESCRIPTION:
Some people have problems with self-assertiveness. That can have negative impact on their lives. This study will test a constructive self-assertiveness intervention program delivered online. In addition, the relative effect of guidance during the intervention will be investigated.

In a randomized controlled trial three groups will be compared:

1. constructive self-assertiveness with guidance
2. constructive self-assertiveness without guidance
3. Waitlist control

The treatment (and wait) will be 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Human,
* At least 18 years old,
* Able to speak and read Swedish,
* Informed consent.

Exclusion Criteria:

* Severe depression (as defined by a PHQ9 score of 15 points or higher),
* If on medication the dosage has been stable for at least the past 3 months,
* No ongoing psychotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-05-16 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Adaptive and Aggressive Assertiveness Scale | Up to 12 months
  A self-report questionnaire measuring Adaptive and Aggressive Assertiveness. Higher scores mean a worse outcome. Minimum and maximum values: 30-150.

SECONDARY OUTCOMES:
Patient Health Questionnaire 9-item | Up to 12 months
  Depression questionnaire. Higher scores mean a worse outcome. Higher scores mean a worse outcome. Minimum and maximum values: 0-27.
Generalized Anxiety Disorder 7 | Up to 12 months
  General Anxiety questionnaire. Higher scores mean a worse outcome. Minimum and maximum values: 0-27.
Liebowitz Social Anxiety Scale , self-report | Up to 12 months
  Social Anxiety questionnaire. Higher scores mean a worse outcome. Minimum and maximum values: 0-144.
Rathus Assertiveness Schedule | Up to 12 months
  Assertiveness questionnaire. Higher scores mean a worse outcome. Minimum and maximum values: -30 to +30.
Well-being scale | Up to 12 months
  Depression scale. Lower scores mean a worse outcome. Minimum and maximum values: 0-72.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Analytic code and pseudoanonymous data in a data repository.
Supporting Information: Analytic Code

REFERENCES:
- [Result] Hagberg T, Manhem P, Oscarsson M, Michel F, Andersson G, Carlbring P. Efficacy of transdiagnostic cognitive-behavioral therapy for assertiveness: A randomized controlled trial. Internet Interv. 2023 May 13;32:100629. doi: 10.1016/j.invent.2023.100629. eCollection 2023 Apr. PMID 37273933
- Available data/document: Individual Participant Data Set — https://github.com/hmep/r2fu/
- Available data/document: Analytic Code — https://github.com/hmep/r2fu/